CLINICAL TRIAL: NCT02449668
Title: Acupuncture Treatment of Shoulder Impingement Syndrome: a Randomized Controlled Trial
Brief Title: Acupuncture Treatment of Shoulder Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rueda, Juan Carlos, M.D., Ph.D. (Individual)
Responsible Party: Principal Investigator, JUAN CARLOS RUEDA GARRIDO, Medical Director, Rueda, Juan Carlos, M.D., Ph.D.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10952-1095
Record Dates: First submitted 2015-05-10; First posted 2015-05-20 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Shoulder Pain
Keywords: Acupuncture; Shoulder pain; Impingement syndrome; Rotator cuff tendinitis; Traditional Chinese medicine (TCM)
MeSH Terms: conditions — Shoulder Pain; Rotator Cuff Injuries | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture on sham points (SA) (Sham Comparator): The control group received treatment with acupuncture needles on sham points (SA).
  Interventions: Device: Sham Acupuncture
- True acupuncture (TA) (Experimental): The intervention group received treatment with true acupuncture techniques (TA) on a selection of points described as effective in the literature.
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — Acupuncture techniques with a plastic insertion tube was used to introduce every needle. The needles were perpendicularly inserted to a depth of 2-3 cm. The needles were applied to the area of the injured shoulder while the patient was lying in a lateral decubitus position on the stretcher. The skin was prepared with clorhexidine and the needles were sterile. They measured 40 mm long and 0.25 mm in diameter. The sessions lasted 20 minutes and the Qi sensation was sought by consistent manipulations, with rotation of the needles in both senses and scratching of the handle.
  Arms: True acupuncture (TA)
Device: Sham Acupuncture
  Arms: Acupuncture on sham points (SA)

SUMMARY:
The main objective of the current study was to assess the analgesic effect achieved to short- and medium-term by the use of acupuncture on individuals with impingement syndrome of the shoulder, in comparison to the use of acupuncture at sham points. Furthermore, secondary objectives were also sought, such as the short- to medium-term functional recovery of the affected joint, knowing the possible influence that this has over the recovery of the laterality of the subject, as well as the development of a protocol to select points to treat pain affecting the shoulder area.

DETAILED DESCRIPTION:
A prospective, controlled, randomized study was carried out. Two parallel, randomly separated groups were monitored. The intervention group received treatment with true acupuncture techniques (TA) on a selection of points described as effective in the literature, and the control group received treatment with acupuncture needles on sham points (SA).

The study was carried out with volunteers, who were informed about its rationale and invited to participate provided they met the following inclusion criteria: they had been diagnosed with the impingement syndrome, with compatible clinical symptoms of more than 3 months of progression; they presented with a unilateral injury; and they had signed their informed consent. Furthermore, the following exclusion criteria were also applied: previous surgery of the injured shoulder; previous luxation or fracture; neurological injuries or illnesses with musculoskeletal disorders.

All the participants who met the selection criteria were invited to an initial consultation to receive information about the study and sign consent. Each participant was randomly assigned to one of the two groups to receive a treatment with: 1) acupuncture at true local and distal points (TA) or 2) acupuncture at sham points (SA).

The random assignment of each participant to one of the two groups of the study was completed when the subjects agreed to participate and signed their consent. Each of them received a code that assigned them to one of the two groups.

The distribution of the participants in each group was also known to the main researcher, having been completed according to a random sequence of codes generated by a random generator program (Numbers®) which produced a list of values (0=acupuncture on sham points (SA); 1=true acupuncture (TA)). Each patient who joined the study received an identification number dictated by the order of their recruitment to the sample, which was matched to the list to include them in one or other of the two groups.

Each participant was informed about the sort of study they were taking part in, but they remained blind to their treatment arm at all times, during both the intervention phase and the monitoring phase.

Each participant received four acupuncture sessions, one per week. Each patient was assessed by one of the researchers in their first consultation before receiving any acupuncture session to obtain a baseline (T0), once the four treatment sessions were completed (T1) and 3 months after the end of the treatment (T2).

After examination of the existing literature, it was decided that an improvement in the perception of pain measured by the VAS (Visual Analogic Scale) of at least a decrease of 20 mm should represent achievement of a clinically significant outcome. In order to obtain a level of significance of 5% and a statistical power of 90%, it was calculated that 62 subjects had to be included in the study. After factoring in an estimated drop-out rate of 10%, a sample of 70 subjects was decided upon.

ELIGIBILITY:
Inclusion Criteria:

* they had been diagnosed with the impingement syndrome
* compatible clinical symptoms of more than 3 months of progression
* they presented with a unilateral injury
* they had signed their informed consent.

Exclusion Criteria:

* previous surgery of the injured shoulder
* previous luxation or fracture
* neurological injuries
* illnesses with musculoskeletal disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Change from baseline in Visual Analogue Scale (VAS) at 3 months after the last session of acupuncture (identified like T2).
  A 100 mm long horizontal bar Visual Analogue Scale (VAS), indicating a maximum and a minimum level of pain in every endpoint. This was used without any other data that could give information to the patient, so that it was presented as a horizontal masked bar.

SECONDARY OUTCOMES:
The Questionnaire of Functional Assessment of the Shoulder, University California (UCLA) | Change from baseline in Questionnaire of Functional Assessment of the Shoulder (UCLA Scale) at 3 months after the last session of acupuncture (identified like T2).
  A brief questionnaire for the functional assessment of the shoulder in general terms[15] which considers 34-35 points as an excellent outcome, 33-28 points a good outcome, 27-21 a medium outcome and 20-0 as a bad outcome.

REFERENCES:
- See also: Trial´s abstract of Doctoral Thesis — http://hdl.handle.net/10952/1095